CLINICAL TRIAL: NCT02061930
Title: Evaluation of the Soft Tissue Stability Around Single Crowns Supported by Tissue Level Implants Placed in Non-augmented Healed Sites in the Anterior Maxilla: a Retrospective Study
Brief Title: Evaluation of the Aesthetic Outcomes of the Single Crowns Supported by Tissue Level Implants
Acronym: PES/WES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Hongchang Lai, Dept. Oral & Maxillofacial Implantology, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: Shanghai9
Record Dates: First submitted 2014-02-07; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Poor Aesthetics of Existing Restoration
Keywords: single tooth; dental implant; aesthetics outcome; long term; soft tissue recession; pink esthetic score; white esthetic score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single crowns supported by implants: single crowns supported by implants placed in the anterior maxilla region, periodontally healthy
  Interventions: Procedure: single crowns supported by implants

INTERVENTIONS:
Procedure: single crowns supported by implants — The implant placement procedures were planned based on clinical and radiographic evaluation. During the surgeries, the mid-crestal incision and intra-crevicular incision were made following local articaine infiltration anesthesia. No releasing incisions were made. After full-thickness flaps were elevated labially and lingually to expose the alveolar ridge, the implants were placed according to the standard surgical procedures defined by the manufacturer. After a healing time of 10-16 weeks, implant-level impressions were taken. The porcelain (Ivoclar-Vivadent AG, Schaan, Lichtenstein) fused to noble metal crowns were fabricated. Abutment screws were torqued to 15 Ncm. Crowns were cemented with HY-bond Glassionomer Cement
  Other Names: Straumann dental implants SLA sp

SUMMARY:
The aim of this study is to review the long-term soft tissue stability and the long-term esthetic results of single crowns supported by tissue level implants placed in non-augmented healed sites.

The hypothesis of the present study is that tissue level implants can achieve ideal esthetic outcomes in non-augmented healed sites.

DETAILED DESCRIPTION:
Both successful implant-supported restorations and the peri-implant soft and hard tissues are vital determinants which may affect the short- and long-term aesthetic outcomes.

For this reason, the pink aesthetic score (PES) was introduced for the evaluation of peri-implant soft tissues by Fürhauser in 2005 and modified by Belser as PES/WES in 2009.

So far, a series of clinical studies have confirmed the suitability of PES/WES and PES index for the objective outcome assessment of the aesthetic dimension of anterior single-tooth implants.

However, to our knowledge, studies with long term data of the aesthetic outcome evaluation in non-augmented healed sites of the anterior maxilla are still rare, for most of the papers published recently mainly focused on immediate implant placement after tooth extraction with only 1-5 years following up.

In our previous study, we have evaluated the alterations of soft tissue around implant-supported single crowns in the anterior maxilla with original standard PES at the time of crown placement and 6 months post-loading .We have found that the aesthetic outcome of soft tissue around the single-tooth implant had improved significantly at follow-up compared with baseline according to PES assessment. However, the follow up time of the previous study was short (6-8 months), long time follow up is necessary to confirm the previous hypothesis and observations.

ELIGIBILITY:
Inclusion Criteria:

* Have had the tooth extraction at least 3 months before implant surgery.
* Did not receive soft or hard tissue augmentation before or in conjunction with implant surgery.
* Did not receive restorative treatment of the adjacent teeth.
* Underwent conventional healing and loading protocol after implant surgery.
* Have both neighboring teeth and corresponding teeth in the mandible.

  ----For additional, the patients should have
* Photographs of the anterior teeth, the photos should have been taken at right after crown placement and at the 6-10 months recall visit.
* Radiographs of the implant-supported single crowns, the radiographs should have been taken at right after crown placement.

Exclusion Criteria:

* Patients who don't fulfill the inclusion criteria
* Patients who refused to join the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Have at least one implant-supported single crown in the anterior maxilla region (13-23) with Straumann (Institute Straumann AG, Waldenburg, Switzerland) tissue level implants placed between December 2005 and October 2008.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
aesthetic scores | baseline
  The photos were taken 1 hour after cementation of the crowns Digital camera will being used during the examinations (Nikon D70, Nikon Medical Objective circular flash; Nikon Corporation, Tokyo, Japan).
  The evaluation will be based on the pictures of the prosthesis and soft tissue around the crown which supported by implant.
  7 parameters will be assessed for PES :mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture.
  5 parameters will be assessed for WES:general tooth form; outline and volume of the clinical crown; color; surface texture; and translucency and characterization.
  For both PES and WES, the score of 2, 1, or 0 is assigned to each parameter by certain evaluation standard
aesthetic scores | 6-10 months after crown placement
  The pictures were taken routinely during patients's revisit . The PES will be assessed via photographs, in order to evaluate the changes of the soft tissue around the crown.
  WES will not be evaluated at this time point.
aesthetic scores | 5-8 years after crown placement
  The photos will be taken by the same digital camera (Nikon D70, Nikon Medical Objective circular flash; Nikon Corporation, Tokyo, Japan)
  both PES and WES will be evaluated at this time point

SECONDARY OUTCOMES:
Modified plaque index (mPLI) | 5-8 years after restoration
  The mPLI will be recorded at four sites (mesial, distal, buccal and palatal) around each of the implant-supported single crowns by a periodontal probe (15 UNC/CP-11.5B Screening Color-Coded Probe
  , Hu-Friedy).
marginal bone resorption | 5-8 years after restoration
  As routine postoperative examination, peri-apical radiographs were taken for all the patients with the long-cone technique at the time when the crowns were cemented. And the latest radiographs will be taken at the time of the last revisit. All of the radiographic films were scanned at 600 dpi with a scanner and the marginal bone level will be assessed with image analysis software.The distance between implant shoulder and first visible bone-to-implant contact (BID) will be measured on the mesial and distal aspects. For each implant and each examination period, the values will be calculated as the average of the obtained mesial and distal values.
Modified sulcus bleeding index (mSBI) | 5-8 years after crown placement
  mSBI will recorded at four sites (mesial, distal, buccal and palatal) around each of the implant-supported single crowns by a periodontal probe (15 UNC/CP-11.5B Screening Color-Coded Probe, Hu-Friedy)
probing depth (PD) | 5-8 years after crown placement
  The peri-implant probing depth was recorded by a periodontal probe (15 UNC/CP-11.5B Screening Color-Coded Probe
  , Hu-Friedy) at the four sites too (Mesial, Distal, buccal, lingual). The recordings were made to the nearest millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Hongchang Lai, DDS, Study Director — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Dept. Oral & Maxillofacial Implantology ,Shanghai 9th People's Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Belser U, Buser D, Higginbottom F. Consensus statements and recommended clinical procedures regarding esthetics in implant dentistry. Int J Oral Maxillofac Implants. 2004;19 Suppl:73-4. No abstract available. PMID 15635947
- [Background] Belser UC, Grutter L, Vailati F, Bornstein MM, Weber HP, Buser D. Outcome evaluation of early placed maxillary anterior single-tooth implants using objective esthetic criteria: a cross-sectional, retrospective study in 45 patients with a 2- to 4-year follow-up using pink and white esthetic scores. J Periodontol. 2009 Jan;80(1):140-51. doi: 10.1902/jop.2009.080435. PMID 19228100
- [Background] Buser D, Chappuis V, Bornstein MM, Wittneben JG, Frei M, Belser UC. Long-term stability of contour augmentation with early implant placement following single tooth extraction in the esthetic zone: a prospective, cross-sectional study in 41 patients with a 5- to 9-year follow-up. J Periodontol. 2013 Nov;84(11):1517-27. doi: 10.1902/jop.2013.120635. Epub 2013 Jan 24. PMID 23347346
- [Background] Grunder U, Gracis S, Capelli M. Influence of the 3-D bone-to-implant relationship on esthetics. Int J Periodontics Restorative Dent. 2005 Apr;25(2):113-9. PMID 15839587
- [Background] Henriksson K, Jemt T. Measurements of soft tissue volume in association with single-implant restorations: a 1-year comparative study after abutment connection surgery. Clin Implant Dent Relat Res. 2004;6(4):181-9. doi: 10.1111/j.1708-8208.2004.tb00034.x. PMID 15841578
- [Background] Cosyn J, Eghbali A, De Bruyn H, Collys K, Cleymaet R, De Rouck T. Immediate single-tooth implants in the anterior maxilla: 3-year results of a case series on hard and soft tissue response and aesthetics. J Clin Periodontol. 2011 Aug;38(8):746-53. doi: 10.1111/j.1600-051X.2011.01748.x. PMID 21752044
- [Background] Cosyn J, Eghbali A, De Bruyn H, Dierens M, De Rouck T. Single implant treatment in healing versus healed sites of the anterior maxilla: an aesthetic evaluation. Clin Implant Dent Relat Res. 2012 Aug;14(4):517-26. doi: 10.1111/j.1708-8208.2010.00300.x. Epub 2010 Jul 17. PMID 20662859
- [Result] Lai HC, Zhang ZY, Wang F, Zhuang LF, Liu X, Pu YP. Evaluation of soft-tissue alteration around implant-supported single-tooth restoration in the anterior maxilla: the pink esthetic score. Clin Oral Implants Res. 2008 Jun;19(6):560-4. doi: 10.1111/j.1600-0501.2008.01522.x. PMID 18474062
- [Result] Meijer HJ, Stellingsma K, Meijndert L, Raghoebar GM. A new index for rating aesthetics of implant-supported single crowns and adjacent soft tissues--the Implant Crown Aesthetic Index. Clin Oral Implants Res. 2005 Dec;16(6):645-9. doi: 10.1111/j.1600-0501.2005.01128.x. PMID 16307570
- [Result] Gallucci GO, Grutter L, Nedir R, Bischof M, Belser UC. Esthetic outcomes with porcelain-fused-to-ceramic and all-ceramic single-implant crowns: a randomized clinical trial. Clin Oral Implants Res. 2011 Jan;22(1):62-9. doi: 10.1111/j.1600-0501.2010.01997.x. Epub 2010 Sep 24. PMID 21158931
- [Result] Dierens M, de Bruecker E, Vandeweghe S, Kisch J, de Bruyn H, Cosyn J. Alterations in soft tissue levels and aesthetics over a 16-22 year period following single implant treatment in periodontally-healthy patients: a retrospective case series. J Clin Periodontol. 2013 Mar;40(3):311-8. doi: 10.1111/jcpe.12049. Epub 2013 Jan 9. PMID 23297745